CLINICAL TRIAL: NCT04426760
Title: Mechanisms of Reduced Fertility in Women With Uterine Leiomyomas
Brief Title: Fibroids and Infertility - a Study of the Significance of Removal of Fibroids With Regard to Endometrial Receptivity
Acronym: FIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kirsten Hald, MD, PhD, Senior Consultant, Oslo University Hospital
Other Study IDs: 2017/9703
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Leiomyoma, Uterine
Keywords: Infertility; Endometrial receptivity; Leiomyoma; Fibroid
MeSH Terms: conditions — Leiomyoma; Infertility | interventions — Laparotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Endometrial biopsies Leiomyoma biopsy Serum Plasma Blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Women with submucosal leiomyoma(s): Women with submucosal leimyomas undergoing hysteroscopical removal of the leiomyoma
  Interventions: Procedure: Transcervical resection of fibroids
- Women with intramural leiomyomas: Women with intramural leiomyomas undergoing myomectomy
  Interventions: Procedure: Myomectomy per laparoscopy or laparotomy
- Infertility patients: Patients treated at the Department for Reproductive Medicine at the Oslo University hospital failing to conceive after 3 or more embryo transfers with good quality embryos.
- Fertile women: Healthy, volunteering women with proved fertility with 1 or more deliveries and no history of infertility

INTERVENTIONS:
Procedure: Transcervical resection of fibroids — Transcervical resection of fibroids
  Groups: Women with submucosal leiomyoma(s)
Procedure: Myomectomy per laparoscopy or laparotomy — Myomectomy per laparoscopy or laparotomy
  Groups: Women with intramural leiomyomas

SUMMARY:
We aim to explore some of the molecular factors that reduce fertility for women with leiomyomas, taking into account leiomyoma location, size, number and vascularity. Tissue samples from the endometrium and leiomyomas will be obtained during the mid secretory phase before and 3-6 months after surgical excision for a comprehensive search for key molecular derangements.

DETAILED DESCRIPTION:
Baseline medical information and standard questionnaire to record symptoms are collected from all participants and a gynaecological examination and a 2D and 3D vaginal ultrasonography including saline infusion sonography (SIS), if indicated, are performed. Blood samples for the biobank for extraction of germ line DNA and for identification of possible biomarkers are taken.

The women with submucosal leiomyomas will undergo hysteroscopic myomectomy and the women with intramural leiomyomas will undergo myomectomy per laparoscopy or laparotomy.

For the participants with intramural leiomyomas and the fertile/infertile controls, endometrial samples are taken with an endometrial suction curette in an outpatient setting at day 19-23 of the menstrual cycle. The endometrial sampling in the group of women with submucosal leiomyomas is being done during the hysteroscopic removal of the leiomyoma, also at day 19-23 of the menstrual cycle.

3-6 months after surgery, cycle day 19-23, endometrial samples will be taken from the women who have undergone myomectomy and ultrasound examination is being performed. The women with submucosal leiomyomas will undergo a second look hysteroscopy

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years
* Presence of leiomyoma(s)
* Regular menstrual cycle (28 +/- 7 days)
* Having had at least 2 normal menstrual cycles after ending the treatment if previously treated with GnRH analogue
* Signed informed consent

Exclusion Criteria:

* No treatment indication (no symptoms and/or no desire for fertility)
* Contraindication for surgery
* Known endometriosis
* Known PCOS
* Untreated hydrosalpinx
* Malignancy; gynaecological or other location
* Pre-malignant or malignant pap smear or endometrial biopsy
* Hormonal treatment including ulipristal acetat and levonorgestrel intrauterine device last three months before inclusion in the study
* Ongoing treatment with GnRH analogue
* Pregnancy last 3 months
* Ongoing lactation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The biological sex must be female since we are studying a phenomenone occuring in the female genital tract.
Study Population: Patients referred to the Department of Gynaecology at Oslo University Hospital for treatment of submucosal or intramural leiomyomas.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
HOXA 10 expression | 3-6 months
  Fold change of HOXA 10 Expression 3-6 months after myomectomy compared to pre-surgery Levels

SECONDARY OUTCOMES:
Expression of other molecular markers | 3-6 months
  Fold change of other molecular markers than HOXA 10 of endometrial receptivity 3-6 months after myomectomy and compared to fertile/infertile controls
Endometrial vascular pattern | 3-6 months
  VI and FI of the endometrium and subendometrial myometrium of women with leimyomas 3-6 months after myomectomy and compared to fertile/infertile controls
Vascular characteristics of leiomyomas | 3-6 months
  Vascular characteristics of leiomyomas associated with endometrial changes
Leiomyoma size | 3-6 months
  Leiomyomas size in centimeters associated with endometrial changes
Leiomyoma location | 3-6 months
  Leiomyoma location associated with endometrial changes
Genomic characteristics | 3-6 months
  Genomic characteristics of leiomyomas associated with endometrial changes
Scar formation | 3-6 months
  Scar/fibrosis/adhesion formation after myomectomy; macroscopically and histologically
Pregnancy | 2 years
  Pregnancy and deliveries within 2 years after myomectomy.
HOXA10 in endometrium of women with leiomyomas compared to fertile/infertile controls | 3-6 months
  Difference in HOXA 10 expression in endometrium of women with leiomyomas compared to fertile/infertile controls
Expression of molecular markers adjacent to the leiomyoma versus remote from the leiomyoma | 3-6 months
  Difference in expression of molecular markers in endometrium adjacent to the leiomyoma compared to endometrium remote from the leiomyoma.
Partially resected leiomyomas | 3-6 months
  Alterations in molecular markers of endometrial receptivity after partially resected submucosal leiomyomas.
Submucosal leiomyomas versus intramural leiomyomas | 3-6 months
  Difference in expression of molecular markers in endometrium of women with submucosal leiomyomas compared with endometrium in women with intramural leiomyomas.
Biomarkers in blood | 1 year
  Biomarkers in blood related to leiomyomas and a possible correlation between certain biomarkers and reduced endometrial receptivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway